CLINICAL TRIAL: NCT02702609
Title: Prospective, Comparative Assessment of Alveolar Ridge Preservation Using GUIDOR® Easy-graft® Classic in Atraumatic Extraction Socket
Brief Title: Assessment of Ridge Preservation Using Moldable Beta-tricalcium Phosphate Bone Grafting System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLP-2015-12-17-1
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Dental Implants; Alveolar Ridge Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moldable beta-TCP grafting system (Experimental): Device: easy-graft CLASSIC (beta-Tricalcium Phosphate)
  Interventions: Device: easy-graft CLASSIC
- Allograft (Active Comparator): Device: Freeze-Dried Bone Allograft (FDBA) with collagen plug
  Interventions: Device: FDBA with collagen plug

INTERVENTIONS:
Device: easy-graft CLASSIC — easy-graft will be grafted to a single extraction socket to preserve the ridge dimension for future implant placement.
  Arms: Moldable beta-TCP grafting system
Device: FDBA with collagen plug — FDBA will be grafted to a single extraction socket and covered by collagen plug to preserve the ridge dimension for future implant placement.
  Arms: Allograft

SUMMARY:
Randomized Controlled study to compare the effectiveness of two different treatment approaches using a new moldable beta-tricalcium phosphate(TCP) bone graft material in ridge preservation of an atraumatic extraction socket site compared to allograft with collagen plug.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* At least 18 years old
* In need of one posterior tooth, excluding third molar molars, planned for extraction and replacement with a dental implant (If the subject requires two adjacent socket preservation, they can still be enrolled in the study but only one site will be used for the study)
* Intact ridge as verified with cone-beam CT scan
* At least one natural tooth adjacent to the study site present.

Exclusion Criteria:

* Insufficient interocclusal space to allow for implant supported prosthesis
* Dehiscence or fenestration identified at the time of reviewing CBCT.
* Non-treated caries or uncontrolled periodontal disease present affecting the teeth in adjacent to study teeth.
* Any of natural teeth adjacent to the study site presents active periapical endodontic lesion ("active periapical endodontic lesion" will be determined per consultation by endodontics specialist).
* Adjacent tooth (mesial and distal) to study site was extracted within last 6 months
* Adjacent teeth (or tooth) to study site with significant soft tissue loss
* Smoker using more than 10 cigarettes or equivalent per day
* Smokeless tobacco use or e-cigarette use
* Current alcohol or drug abuser
* Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration e.g. uncontrolled diabetes
* Need for systemic corticosteroids or any other medication that would influence post-operative healing and/or osseointegration
* Pregnancy, as indicated by positive serum human chorionic gonadotropin (HCG) test result.
* Unable or unwilling to return for follow-up visits for a period of 5 months
* Unlikely to be able to comply with study procedures according to Investigators judgement
* Subject in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Iowa College of Dentistry, Iowa City, Iowa
  - University of Maryland School of Dentistry, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled at 2 dental schools between August 2016 and June 2017.
Period: Overall Study
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Started | 24 | 21
Implant Placement | 23 | 21
Crown Delivery | 16 | 18
Completed | 15 | 17
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 8 | 4
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moldable Beta-TCP Grafting System | Allograft | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.2) | 53.5 (11.4) | 57.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 20 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 22 | 16 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking history [Count of Participants; unit: Participants]
  Smoker | 1 | 2 | 3
  Non-smoker | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Radiographic Measurements of Ridge Dimension (Horizontal Ridge Width)
Description: Cone-beam computed tomography (CBCT) is taken at the ridge preservation procedure (baseline) and 4 months after the procedure. Linear measurement of horizontal ridge width is measured at 1 mm apical to the crest. Change of horizontal ridge width = (Baseline measurement - 4 months measurement)
Time Frame: Baseline and 4 months post-surgery
Population: The modified Intent-to-Treat population consisted of 43 subjects after a subject was removed for lack of compliance with the study protocol.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Number analyzed (Participants) | 23 | 20
mm | 1.26 (1.32) | 1.28 (1.73)

2. Primary Outcome: Change in Radiographic Measurements of Ridge Dimension (Volumetric Assessment)
Description: Cone-beam computed tomography (CBCT) is taken at the ridge preservation procedure (baseline) and 4 months after the procedure. Bone volume measurement is expressed in mm3, which allowed for a calculation of the % of volumetric reduction that took place from baseline to 4 months post-surgery.
Time Frame: Baseline and 4 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of volume at baseline
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Number analyzed (Participants) | 23 | 20
percentage of volume at baseline | 23.9 (22.1) | 17.0 (15.4)

3. Secondary Outcome: Histomorphometric Assessment of Newly Formed Mineralized Tissue
Description: Bone core biopsy is harvested at the time of implant placement from the "central" part of the ridge at 5 months after ridge preservation procedure. Histomorphometric analysis is performed by one blinded examiner who measured a proportion of mineralized tissue respective to the percent of the total core area.
Time Frame: 5 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total core area
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Number analyzed (Participants) | 23 | 20
percentage of total core area | 27.0 (22.1) | 38.2 (12.5)

4. Secondary Outcome: Histomorphometric Assessment of Residual Bone Graft Particles
Description: Bone core biopsy is harvested at the time of implant placement from the "central" part of the ridge at 5 months after ridge preservation procedure. Histomorphometric analysis is performed by one blinded examiner who measured a proportion of residual bone graft respective to the percent of the total core area.
Time Frame: 5 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total core area
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Number analyzed (Participants) | 23 | 20
percentage of total core area | 20.5 (16.8) | 15.7 (7.0)

5. Secondary Outcome: Histomorphometric Assessment of Non-mineralized Tissue
Description: Bone core biopsy is harvested at the time of implant placement from the "central" part of the ridge at 5 months after ridge preservation procedure. Histomorphometric analysis is performed by one blinded examiner who measured a proportion of non-mineralized tissue respective to the percent of the total core area.
Time Frame: 5 months post-surgery
Measure: Mean (Standard Deviation); unit: percentage of total core area
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Number analyzed (Participants) | 23 | 20
percentage of total core area | 52.5 (11.8) | 46.1 (10.5)

6. Secondary Outcome: Change of Marginal Bone Level Around Dental Implant
Description: Linear measurement of marginal bone level (MBL) in millimeters along mesial and distal dental implant surface are captured in periapical standardized radiographs at crown delivery (baseline), 6, and 12 months after crown delivery. Change of MBL = (Baseline measurement - 6 or 12 months measurement)
Time Frame: Baseline, 6, and 12 months after crown delivery
Population: 34 subjects received crown delivery on the study site after implant placement and two subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
Number analyzed (Participants) | 15 | 17
mm
  Mesial 6 months | 0.04 (0.06) | 0.06 (0.07)
  Distal 6 months | 0.12 (0.05) | -0.05 (0.06)
  Mesial 12 months | 0.02 (0.07) | 0.02 (0.09)
  Distal 12 months | 0.09 (0.08) | 0.09 (0.07)

ADVERSE EVENTS:
Time Frame: One year after crown delivery
Arm/Group | Moldable Beta-TCP Grafting System | Allograft
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 2/24 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moldable Beta-TCP Grafting System (N=24) | Allograft (N=21)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1)
Oroantral fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — Preexisting condition was updated.
Dental restoration failure (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will submit the manuscript of the proposed publication or presentation to Sponsor at least 30 days prior to publication or release, or submission for the publication of any manuscript, and Sponsor shall have the right to review and comment upon the publication in order to protect Sponsor's confidential information. Upon Sponsor's written request, publication will be delayed up to 60 additional days to enable Sponsor to secure adequate intellectual property protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02702609/Prot_SAP_000.pdf